CLINICAL TRIAL: NCT01429974
Title: Detection of Meconium in Amniotic Fluid in Post Term Pregnancies
Status: Terminated | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-11-8479-AO-CTIL
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Meconium
Keywords: amniotic fluid; post term pregnancies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- volunteers
  Interventions: Other: amniometer model po1

INTERVENTIONS:
Other: amniometer model po1 — The detection of Meconium, is based on recognizing a characteristic fluoroscopic spectral pattern emitted by Meconium under light excitation at a specific wavelength.
  The diagnostic test does not require penetration into the amniotic sac and is safe, painless and simple to perform.

SUMMARY:
Meconium constitutes the bowel contents of the fetus and is normally expelled only after birth. However, it may be secreted into the amniotic fluid of 20% of all fetuses. Meconium Stained Amniotic Fluid had been recognized from ancient times as an obstetric hazard which complicates delivery and is associated with increased newborn morbidity and mortality. At present there is no viable diagnostic test for Meconium prior to the onset of labor and the rupture of membranes. The system developed for the detection of Meconium, based on recognizing a characteristic fluoroscopic spectral pattern emitted by Meconium under light excitation at a specific wavelength. The diagnostic test being developed does not require penetration into the amniotic sac and is safe, painless and simple to perform.

ELIGIBILITY:
Inclusion Criteria:

* 37-42 weeks regnancy without rupture of membranes

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post term pregnant females
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
Determine the capability for diagnosing Meconium stained Amniotic Fluid prior to a cervical ripening procedure in women, using the Amniometer device | prior to breakage of water

CONTACTS AND LOCATIONS:
Overall Officials: Arie Orenstein, professor, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel